CLINICAL TRIAL: NCT03965962
Title: Immunogenicity and Safety of a Purified Vero Rabies Vaccine - Serum Free in Comparison With Verorab® and Imovax® Rabies, in a Simulated Rabies Post-exposure Regimen in Healthy Adults in France
Brief Title: Study of Purified Vero Rabies Vaccine Compared With Two Reference Rabies Vaccines in a Simulated Post-Exposure Regimen in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VRV13; 2018-004055-20 (EudraCT Number); U1111-1216-6151 (Other: UTN)
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Rabies (Healthy Volunteers)
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Intervention Model Description: The study was divided into 4 groups: groups 1 to 3 (VRVg-2 + HRIG; Verorab + HRIG; Imovax Rabies + HRIG) were modified double-blind and group 4 (VRVg-2 standalone) was open-label.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind: the participant (or legally acceptable representative) and the Investigator remain unaware of the treatment assignments throughout the study. An unblinded qualified trial staff member administered the appropriate vaccine but was not involved in the immunogenicity and safety evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: VRVg-2 + HRIG (Experimental): Participants received 0.5 milliliters (mL) intramuscular (IM) injection of VRVg-2 formulation on Days 0, 3, 7, 14 and 28 along with HRIG injection at Day 0.
  Interventions: Biological: VRVg-2; Biological: Rabies immune globulin (human)
- Group 2: Verorab + HRIG (Active Comparator): Participants received 0.5 mL IM injection of Verorab on Days 0, 3, 7, 14 and 28 along with HRIG injection at Day 0.
  Interventions: Biological: Purified Inactivated Rabies Vaccine; Biological: Rabies immune globulin (human)
- Group 3: Imovax Rabies + HRIG (Active Comparator): Participants received 1 mL IM injection of Imovax Rabies on Days 0, 3, 7, 14 and 28 along with HRIG injection at Day 0.
  Interventions: Biological: Human Diploid Cell Vaccine (HDCV); Biological: Rabies immune globulin (human)
- Group 4: VRVg-2 (Experimental): Participants received 0.5 mL IM injection of VRVg-2 formulation on Days 0, 3, 7, 14 and 28.
  Interventions: Biological: VRVg-2

INTERVENTIONS:
Biological: VRVg-2 — Pharmaceutical form: Powder and solvent for suspension for injection;
  Route of administration: IM
  Arms: Group 1: VRVg-2 + HRIG; Group 4: VRVg-2
Biological: Purified Inactivated Rabies Vaccine — Pharmaceutical form: Powder and solvent for suspension for injection;
  Route of administration: IM
  Other Names: Verorab®
  Arms: Group 2: Verorab + HRIG
Biological: Human Diploid Cell Vaccine (HDCV) — Pharmaceutical form: Powder and solvent for suspension for injection;
  Route of administration: IM
  Other Names: IMOVAX® Rabies
  Arms: Group 3: Imovax Rabies + HRIG
Biological: Rabies immune globulin (human) — Pharmaceutical form: Solution for injection;
  Route of administration: IM
  Other Names: IMOGAM® Rabies-HT
  Arms: Group 1: VRVg-2 + HRIG; Group 2: Verorab + HRIG; Group 3: Imovax Rabies + HRIG

SUMMARY:
Primary Objective:

To demonstrate that Purified Vero Rabies Vaccine - Serum Free Vaccine generation 2 (VRVg-2) was non-inferior to Verorab and Imovax Rabies vaccines when co-administered with human rabies immunoglobulin (HRIG), in terms of proportion of participants achieving a rabies virus neutralizing antibody (RVNA) titer greater than or equal to (>=) 0.5 international units per milliliter (IU/mL) at Day 28, i.e., 14 days after the fourth vaccine injection.

Secondary Objective:

* To describe the safety profile of VRVg-2 versus Verorab and Imovax Rabies vaccines when co-administered with HRIG, as well as that of VRVg-2, after each vaccine injection.
* To demonstrate that the proportion of participants in the VRVg-2 + HRIG group achieving an RVNA titer >= 0.5 IU/mL at Day 28 was at least 95 percent (%).
* To describe the immune response induced by VRVg-2 versus Verorab and Imovax Rabies vaccines when co-administered with HRIG, as well as that induced by VRVg-2, at Day 14 (7 days after the third injection), at Day 28 (14 days after the fourth injection) and at Day 42 (14 days after the last injection).

DETAILED DESCRIPTION:
Study duration per participant was approximately 7 months including: 1 day of screening and vaccination, a total of 5 vaccine injections over a 28-day period, 1 safety-follow up visit at Day 42, 1 safety follow-up/end of study visit at Day 56 and a 6-month safety follow-up call after last vaccine administration.

ELIGIBILITY:
Inclusion criteria :

* Men or women aged >=18 years on the day of inclusion (>= 18 years means from the day of the 18th birthday onwards, with no upper age limit).
* Able to attend all scheduled visits and to comply with all trial procedures.
* Body Mass Index (BMI): 18.5 kilograms per square meter (kg/m^2) less than or equal to (<=) BMI <=30 kg/m^2.

Exclusion criteria:

* Pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile.
* Participation at the time of study enrollment or, planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the first trial vaccination or planned receipt of any vaccine prior to Visit 7.
* Previous vaccination against rabies (in pre- or post-exposure regimen) with either the trial vaccines or another vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* At high risk for rabies exposure during the trial (veterinarians and their staff, animal handlers, rabies researchers, and certain laboratory workers, persons whose activities bring them into frequent contact with rabies virus or potentially rabid bats, raccoons, skunks, cats, dogs, or other species at risk for having rabies, people travelling where rabies was enzootic).
* Known systemic hypersensitivity to any of the vaccine or HRIG components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Self-reported thrombocytopenia, contraindicating IM vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination.
* Current alcohol or substance abuse that, in the opinion of the investigator, might interfere with the trial conduct of completion.
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature >=38.0 degree Celsius). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Personal history of Guillain-Barré syndrome.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (2):
- France (2):
  - Investigational Site Number 2500002, Gières
  - Investigational Site Number 2500001, Rennes

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Pineda-Pena AC, Jiang Q, Petit C, Korejwo-Peyramond J, Donazzolo Y, Latreille M, Homery MC, Babin V, Benamor S, Pichon S, Guinet-Morlot F, Minutello AM. Immunogenicity and Safety of a Purified Vero Rabies Vaccine-Serum Free, Compared With 2 Licensed Vaccines, in a Simulated Rabies Post-Exposure Regimen in Healthy Adults in France: A Randomized, Controlled, Phase 3 Trial. Clin Infect Dis. 2024 Jun 14;78(6):1748-1756. doi: 10.1093/cid/ciae137. PMID 38478634
- See also: VRV13 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25384&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 active centers in France.
Pre-assignment Details: A total of 640 participants were enrolled in the study. Data presented in the disposition table (all milestones) is based on randomized group, except for safety analysis set (SafAS) milestone which is presented based on the actual vaccination group.
Groups:
- Group 1 VRVg-2+HRIG: Participants received 0.5 milliliters (mL) intramuscular (IM) injection of Purified Vero Rabies Vaccine - Serum Free Vaccine generation 2 (VRVg-2) formulation on Days 0, 3, 7, 14 and 28 along with Human Rabies Immunoglobulins (HRIG) injection at Day 0.
- Group 2 Verorab+HRIG: Participants received 0.5 mL IM injection of Verorab on Days 0, 3, 7, 14 and 28 along with HRIG injection at Day 0.
- Group 3 Imovax Rabies+HRIG: Participants received 1 mL IM injection of Imovax Rabies on Days 0, 3, 7, 14 and 28 along with HRIG injection at Day 0.
- Group 4 VRVg-2: Participants received 0.5 mL IM injection of VRVg-2 formulation on Days 0, 3, 7, 14 and 28.
Period: Overall Study
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
Started | 320 | 107 | 107 | 106
Vaccination 1 (Day 0) | 318 | 107 | 107 | 106
Vaccination 2 (Day 3) | 317 | 104 | 107 | 106
Vaccination 3 (Day 7) | 311 | 103 | 105 | 105
Vaccination 4 (Day 14) | 301 | 101 | 101 | 103
Vaccination 5 (Day 28) | 294 | 98 | 97 | 98
Safety Analysis Set (SafAS) (SafAS: Participant who received at least one dose of vaccine and were analyzed as per actual vaccination received.) | 320 (2 participants randomized to Group 4: VRVg-2 received vaccination in Group 1: VRVg-2+HRIG and were considered in Group 1 for safety analysis purpose.) | 107 | 107 | 104 (2 participants randomized to Group 4: VRVg-2 received vaccination in Group 1: VRVg-2+HRIG and were considered in Group 1 for safety analysis purpose.)
Completed | 295 | 102 | 97 | 100
Not Completed | 25 | 5 | 10 | 6
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 21 | 4 | 10 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2 | Total Title
Number analyzed (Participants) | 320 | 107 | 107 | 106 | 640
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (14.7) | 46.2 (14.8) | 46.3 (15.6) | 46.4 (15.0) | 46.1 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 61 | 65 | 60 | 382
  Male | 124 | 46 | 42 | 46 | 258
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 0 | 0 | 4
  Asian | 4 | 1 | 3 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 1 | 0 | 1 | 11
  White | 301 | 102 | 104 | 105 | 612
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 3 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Rabies Virus Neutralizing Antibody (RVNA) Titers Greater Than or Equal to (>=) 0.5 International Units Per Milliliter (IU/mL)-Non-Inferiority Analysis
Description: RVNA titer against rabies virus was assessed using the Rapid Fluorescent Focus Inhibition test (RFFIT) assay method.
Time Frame: Day 28
Population: Analysis was performed on the per-protocol analysis set (PPAS) that included all participants who received at least 1 dose of the study vaccines. The participants who presented protocol deviations, met PPAS exclusion criteria were excluded from PPAS. Data for this outcome measure was planned to be collected and analyzed only for Groups 1, 2, and 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG
Number analyzed (Participants) | 239 | 77 | 78
percentage of participants | 99.6 [97.7 to 100] | 100 [95.3 to 100] | 98.7 [93.1 to 100]
Statistical Analysis 1: Comparison: Group 1 VRVg-2+HRIG vs Group 2 Verorab+HRIG; Test type: Non-Inferiority — The two-sided 95 percent (%) confidence interval (CI) was calculated based on the Wilson score method without continuity correction. Non-inferiority was demonstrated if the lower limit of the 95% CI of the difference of the percentages between the test group (Group 1) and control group (Group 2) was greater than (>) -5% at Day 28; Difference in Percentage = -0.42, 95% CI 2-sided [-2.33 to 4.35]
Statistical Analysis 2: Comparison: Group 1 VRVg-2+HRIG vs Group 3 Imovax Rabies+HRIG; Test type: Non-Inferiority — The two-sided 95 % CI was calculated based on the Wilson score method without continuity correction. Non-inferiority was demonstrated if the lower limit of the 95% CI of the difference of the percentages between the test group (Group 1) and control group (Group 3) was > -5% at Day 28; Difference in Percentage = 0.86, 95% CI 2-sided [-1.32 to 6.50]

2. Secondary Outcome: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.5 IU/mL
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. Immune response of VRVg-2 was considered sufficient if the lower limit of the 95% CI for percentage of participants in Group 1 with RVNA titers >=0.5 IU/mL was not less than 95% at Day 28, when the primary non-inferiority objective was achieved at Day 28.
Time Frame: Day 0 (pre-vaccination), Day 14, Day 28 and Day 42
Population: Analysis was performed on the PPAS. Here, 'number analyzed' signifies participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
Number analyzed (Participants) | 239 | 77 | 78 | 77
percentage of participants
  Day 0 | 0 [0 to 1.5] | 0 [0 to 4.7] | 0 [0 to 4.6] | 0 [0 to 4.7]
  Day 14: number analyzed (Participants) | 213 | 75 | 68 | 69
  Day 14 | 92.5 [88.1 to 95.6] | 88.0 [78.4 to 94.4] | 94.1 [85.6 to 98.4] | 97.1 [89.9 to 99.6]
  Day 28 | 99.6 [97.7 to 100] | 100 [95.3 to 100] | 98.7 [93.1 to 100] | 100 [95.3 to 100]
  Day 42: number analyzed (Participants) | 226 | 74 | 76 | 76
  Day 42 | 100 [98.4 to 100] | 100 [95.1 to 100] | 98.7 [92.9 to 100] | 100 [95.3 to 100]

3. Secondary Outcome: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.2 IU/mL (Lower Limit of Quantification [LLOQ])
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. Lower limit of quantitation (LLOQ) for the RFFIT assay was 0.2 IU/mL.
Time Frame: Day 0 (pre-vaccination), Day 14, Day 28 and Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
Number analyzed (Participants) | 239 | 77 | 78 | 77
percentage of participants
  Day 0 | 0 [0 to 1.5] | 0 [0 to 4.7] | 0 [0 to 4.6] | 0 [0 to 4.7]
  Day 14: number analyzed (Participants) | 213 | 75 | 68 | 69
  Day 14 | 99.5 [97.4 to 100] | 100 [95.2 to 100] | 98.5 [92.1 to 100] | 100 [94.8 to 100]
  Day 28 | 100 [98.5 to 100] | 100 [95.3 to 100] | 98.7 [93.1 to 100] | 100 [95.3 to 100]
  Day 42: number analyzed (Participants) | 226 | 74 | 76 | 76
  Day 42 | 100 [98.4 to 100] | 100 [95.1 to 100] | 100 [95.3 to 100] | 100 [95.3 to 100]

4. Secondary Outcome: Rabies Virus Neutralizing Antibody (RVNA) Geometric Mean Titers (GMTs) Against Rabies Virus
Description: RVNA GMT against rabies virus was assessed using the RFFIT assay method.
Time Frame: Day 0 (pre-vaccination), Day 14, Day 28 and Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
Number analyzed (Participants) | 239 | 77 | 78 | 77
IU/mL
  Day 0 | 0.100 [0.100 to 0.101] | 0.100 [NA to NA] — Upper and lower limits of 95% CI were not estimable because all the participants had same value and no variability was observed. | 0.100 [NA to NA] — Upper and lower limits of 95% CI were not estimable because all the participants had same value and no variability was observed. | 0.101 [0.099 to 0.102]
  Day 14: number analyzed (Participants) | 213 | 75 | 68 | 69
  Day 14 | 2.40 [2.09 to 2.76] | 1.86 [1.44 to 2.41] | 1.83 [1.46 to 2.28] | 5.41 [4.24 to 6.90]
  Day 28 | 6.49 [5.75 to 7.34] | 5.03 [3.94 to 6.44] | 5.51 [4.35 to 6.96] | 12.4 [10.5 to 14.5]
  Day 42: number analyzed (Participants) | 226 | 74 | 76 | 76
  Day 42 | 13.6 [12.3 to 15.0] | 9.47 [7.96 to 11.3] | 10.7 [8.97 to 12.7] | 19.8 [17.5 to 22.5]

5. Secondary Outcome: Geometric Mean Titer Ratio (GMTR) of Rabies Virus Neutralizing Antibody Titers
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. GMTRs were calculated as the ratio of GMTs post vaccination (i.e., on Day 14, 28 and Day 42) and pre-vaccination on Day 0.
Time Frame: Day 0 (pre-vaccination), Day 14, Day 28 and Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
Number analyzed (Participants) | 239 | 77 | 78 | 77
ratio
  Day 14/Day 0: number analyzed (Participants) | 213 | 75 | 68 | 69
  Day 14/Day 0 | 24.0 [20.8 to 27.6] | 18.6 [14.4 to 24.1] | 18.3 [14.6 to 22.8] | 53.7 [42.1 to 68.4]
  Day 28/Day 0 | 64.8 [57.3 to 73.2] | 50.3 [39.4 to 64.4] | 55.1 [43.5 to 69.6] | 123 [105 to 144]
  Day 42/Day 0: number analyzed (Participants) | 226 | 74 | 76 | 76
  Day 42/Day 0 | 135 [122 to 149] | 94.7 [79.6 to 113] | 107 [89.7 to 127] | 197 [173 to 224]

6. Secondary Outcome: Percentage of Participants With Determined Complete and Determined Incomplete Virus Neutralization
Description: Virus neutralization was defined as complete (absence of fluorescent cells) and incomplete (presence of fluorescent cells) at the participant/timepoint level at the starting dilution (1/5) of RFFIT assay. Percentage of participants with determined complete and determined incomplete virus neutralization were reported.
Time Frame: Day 0 (pre-vaccination), Day 14, Day 28 and Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
Number analyzed (Participants) | 239 | 77 | 78 | 77
percentage of participants
  Day 0: Complete Neutralization: number analyzed (Participants) | 231 | 74 | 72 | 74
  Day 0: Complete Neutralization | 0.4 [0 to 2.4] | 0 [0 to 4.9] | 0 [0 to 5.0] | 1.4 [0 to 7.3]
  Day 0: Incomplete Neutralization: number analyzed (Participants) | 231 | 74 | 72 | 74
  Day 0: Incomplete Neutralization | 99.6 [97.6 to 100] | 100 [95.1 to 100] | 100 [95.0 to 100] | 98.6 [92.7 to 100]
  Day 14: Complete Neutralization: number analyzed (Participants) | 229 | 75 | 75 | 77
  Day 14: Complete Neutralization | 98.7 [96.2 to 99.7] | 100 [95.2 to 100] | 98.7 [92.8 to 100] | 98.7 [93.0 to 100]
  Day 14: Incomplete Neutralization: number analyzed (Participants) | 229 | 75 | 75 | 77
  Day 14: Incomplete Neutralization | 1.3 [0.3 to 3.8] | 0 [0 to 4.8] | 1.3 [0 to 7.2] | 1.3 [0 to 7.0]
  Day 28: Complete Neutralization: number analyzed (Participants) | 237 | 77 | 78 | 77
  Day 28: Complete Neutralization | 100 [98.5 to 100] | 100 [95.3 to 100] | 98.7 [93.1 to 100] | 100 [95.3 to 100]
  Day 28: Incomplete Neutralization: number analyzed (Participants) | 237 | 77 | 78 | 77
  Day 28: Incomplete Neutralization | 0 [0 to 1.5] | 0 [0 to 4.7] | 1.3 [0 to 6.9] | 0 [0 to 4.7]
  Day 42: Complete Neutralization: number analyzed (Participants) | 236 | 77 | 78 | 77
  Day 42: Complete Neutralization | 100 [98.4 to 100] | 100 [95.3 to 100] | 100 [95.4 to 100] | 100 [95.3 to 100]
  Day 42: Incomplete Neutralization: number analyzed (Participants) | 236 | 77 | 78 | 77
  Day 42: Incomplete Neutralization | 0 [0 to 1.6] | 0 [0 to 4.7] | 0 [0 to 4.6] | 0 [0 to 4.7]

7. Secondary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study vaccine and does not necessary had to have a causal relationship with treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset post-vaccination. All participants were observed for 30 minutes after any vaccination, and any unsolicited AEs occurred during that time were recorded as immediate unsolicited AEs in the CRB. Immediate AEs considered as related to vaccination were recorded as immediate unsolicited adverse reactions (ARs).
Time Frame: Within 30 minutes after any and each vaccination (Vaccination 1, 2, 3, 4 and 5)
Population: Analysis was performed on the safety analysis set (SafAS) that included participant who had received at least one dose of the study vaccine and were analyzed according to the actual treatment received. Here, 'number analyzed' signifies participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
Number analyzed (Participants) | 320 | 107 | 107 | 104
Participants
  Post-any vaccination | 3 | 0 | 0 | 1
  Post-vaccination 1 | 3 | 0 | 0 | 1
  Post-vaccination 2: number analyzed (Participants) | 319 | 104 | 107 | 104
  Post-vaccination 2 | 0 | 0 | 0 | 0
  Post-vaccination 3: number analyzed (Participants) | 313 | 103 | 105 | 103
  Post-vaccination 3 | 0 | 0 | 0 | 0
  Post-vaccination 4: number analyzed (Participants) | 303 | 101 | 101 | 101
  Post-vaccination 4 | 0 | 0 | 0 | 0
  Post-vaccination 5: number analyzed (Participants) | 296 | 98 | 97 | 96
  Post-vaccination 5 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: A solicited reaction (SR) was an expected AR observed and reported under conditions (nature and onset) prelisted (i.e., solicited) in the protocol and CRB and considered as related to vaccination. An AR was all noxious and unintended responses to a medicinal product related to any dose. Solicited injection site reactions included pain, erythema and swelling at and around the injection site.
Time Frame: Within 7 days after any and each vaccination (Vaccination 1, 2, 3, 4 and 5)
Population: Analysis was performed on the SafAS. Here, 'number analyzed' signifies participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
Number analyzed (Participants) | 320 | 107 | 107 | 104
Participants
  Pain Post-any vaccination | 142 | 37 | 49 | 44
  Pain Post-vaccination 1 | 71 | 19 | 25 | 23
  Pain Post-vaccination 2: number analyzed (Participants) | 319 | 104 | 107 | 104
  Pain Post-vaccination 2 | 84 | 17 | 17 | 20
  Pain Post-vaccination 3: number analyzed (Participants) | 312 | 103 | 105 | 103
  Pain Post-vaccination 3 | 73 | 14 | 23 | 23
  Pain Post-vaccination 4: number analyzed (Participants) | 300 | 101 | 100 | 100
  Pain Post-vaccination 4 | 69 | 12 | 29 | 27
  Pain Post-vaccination 5: number analyzed (Participants) | 295 | 98 | 97 | 96
  Pain Post-vaccination 5 | 40 | 12 | 24 | 21
  Erythema Post-any vaccination | 5 | 5 | 3 | 1
  Erythema Post-vaccination 1 | 0 | 1 | 1 | 0
  Erythema Post-vaccination 2: number analyzed (Participants) | 319 | 104 | 107 | 104
  Erythema Post-vaccination 2 | 0 | 0 | 0 | 0
  Erythema Post-vaccination 3: number analyzed (Participants) | 312 | 103 | 105 | 103
  Erythema Post-vaccination 3 | 0 | 1 | 1 | 0
  Erythema Post-vaccination 4: number analyzed (Participants) | 300 | 101 | 100 | 100
  Erythema Post-vaccination 4 | 3 | 3 | 1 | 1
  Erythema Post-vaccination 5: number analyzed (Participants) | 295 | 98 | 97 | 96
  Erythema Post-vaccination 5 | 2 | 1 | 1 | 0
  Swelling Post-any vaccination | 5 | 1 | 1 | 0
  Swelling Post-vaccination 1 | 1 | 0 | 0 | 0
  Swelling Post-vaccination 2: number analyzed (Participants) | 319 | 104 | 106 | 104
  Swelling Post-vaccination 2 | 0 | 0 | 0 | 0
  Swelling Post-vaccination 3: number analyzed (Participants) | 312 | 103 | 105 | 103
  Swelling Post-vaccination 3 | 2 | 0 | 1 | 0
  Swelling Post-vaccination 4: number analyzed (Participants) | 300 | 101 | 100 | 100
  Swelling Post-vaccination 4 | 2 | 0 | 0 | 0
  Swelling Post-vaccination 5: number analyzed (Participants) | 295 | 98 | 97 | 96
  Swelling Post-vaccination 5 | 1 | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With Solicited Systemic Reactions
Description: SR was an expected AR observed and reported under conditions (nature and onset) prelisted (i.e., solicited) in the protocol and CRB and considered as related to vaccination. An AR was all noxious and unintended responses to a medicinal product related to any dose. Solicited systemic reactions included fever, headache, malaise and myalgia.
Time Frame: Up to 7 days after any and each vaccination (Vaccination 1, 2, 3, 4 and 5)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
Number analyzed (Participants) | 320 | 107 | 107 | 104
Participants
  Fever Post-any vaccination: number analyzed (Participants) | 319 | 107 | 107 | 104
  Fever Post-any vaccination | 4 | 2 | 4 | 1
  Fever Post-vaccination 1: number analyzed (Participants) | 319 | 107 | 107 | 104
  Fever Post-vaccination 1 | 0 | 0 | 1 | 0
  Fever Post-vaccination 2: number analyzed (Participants) | 318 | 104 | 107 | 104
  Fever Post-vaccination 2 | 0 | 0 | 1 | 0
  Fever Post-vaccination 3: number analyzed (Participants) | 311 | 103 | 105 | 103
  Fever Post-vaccination 3 | 2 | 1 | 1 | 0
  Fever Post-vaccination 4: number analyzed (Participants) | 300 | 101 | 100 | 100
  Fever Post-vaccination 4 | 0 | 0 | 2 | 1
  Fever Post-vaccination 5: number analyzed (Participants) | 295 | 97 | 97 | 95
  Fever Post-vaccination 5 | 2 | 1 | 1 | 0
  Headache Post-any vaccination | 107 | 35 | 38 | 36
  Headache Post-vaccination 1 | 44 | 20 | 18 | 17
  Headache Post-vaccination 2: number analyzed (Participants) | 319 | 104 | 107 | 104
  Headache Post-vaccination 2 | 26 | 10 | 10 | 6
  Headache Post-vaccination 3: number analyzed (Participants) | 312 | 103 | 105 | 103
  Headache Post-vaccination 3 | 38 | 13 | 16 | 14
  Headache Post-vaccination 4: number analyzed (Participants) | 300 | 101 | 100 | 100
  Headache Post-vaccination 4 | 29 | 10 | 5 | 14
  Headache Post-vaccination 5: number analyzed (Participants) | 295 | 98 | 97 | 96
  Headache Post-vaccination 5 | 23 | 7 | 5 | 13
  Malaise Post-any vaccination | 34 | 13 | 14 | 13
  Malaise Post-vaccination 1 | 20 | 7 | 5 | 4
  Malaise Post-vaccination 2: number analyzed (Participants) | 319 | 104 | 107 | 104
  Malaise Post-vaccination 2 | 7 | 3 | 5 | 1
  Malaise Post-vaccination 3: number analyzed (Participants) | 312 | 103 | 105 | 103
  Malaise Post-vaccination 3 | 9 | 4 | 4 | 6
  Malaise Post-vaccination 4: number analyzed (Participants) | 300 | 101 | 100 | 100
  Malaise Post-vaccination 4 | 8 | 1 | 1 | 6
  Malaise Post-vaccination 5: number analyzed (Participants) | 295 | 98 | 97 | 96
  Malaise Post-vaccination 5 | 6 | 0 | 2 | 2
  Myalgia Post-any vaccination | 118 | 37 | 38 | 33
  Myalgia Post-vaccination 1 | 58 | 17 | 23 | 20
  Myalgia Post-vaccination 2: number analyzed (Participants) | 319 | 104 | 107 | 104
  Myalgia Post-vaccination 2 | 50 | 11 | 9 | 14
  Myalgia Post-vaccination 3: number analyzed (Participants) | 312 | 103 | 105 | 103
  Myalgia Post-vaccination 3 | 50 | 13 | 15 | 12
  Myalgia Post-vaccination 4: number analyzed (Participants) | 300 | 101 | 100 | 100
  Myalgia Post-vaccination 4 | 35 | 8 | 14 | 17
  Myalgia Post-vaccination 5: number analyzed (Participants) | 295 | 98 | 97 | 96
  Myalgia Post-vaccination 5 | 26 | 8 | 10 | 11

10. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An AE was defined as any untoward medical occurrence in a participant who received study vaccine and does not necessary had to have a causal relationship with treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRB in terms of diagnosis and/or onset post-vaccination.
Time Frame: Up to 28 days after any and each vaccination (Vaccination 1, 2, 3, 4 and 5)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
Number analyzed (Participants) | 320 | 107 | 107 | 104
Participants
  Post-any vaccination | 145 | 46 | 39 | 42
  Post-vaccination 1 | 47 | 22 | 12 | 10
  Post-vaccination 2: number analyzed (Participants) | 319 | 104 | 107 | 104
  Post-vaccination 2 | 27 | 5 | 11 | 5
  Post-vaccination 3: number analyzed (Participants) | 313 | 103 | 105 | 103
  Post-vaccination 3 | 31 | 9 | 7 | 8
  Post-vaccination 4: number analyzed (Participants) | 303 | 101 | 101 | 101
  Post-vaccination 4 | 37 | 9 | 14 | 11
  Post-vaccination 5: number analyzed (Participants) | 296 | 98 | 97 | 96
  Post-vaccination 5 | 60 | 11 | 12 | 21

11. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study vaccine and does not necessary had to have a causal relationship with treatment. An SAE was any untoward medical occurrence that at any dose resulted in death, life-threatening, initial or prolonged inpatient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect or a medically important event. An AESI was defined as one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor was appropriate. All SAEs and AESIs occurring during the study that were related to the product administered were reported by the Investigator to the Independent Ethics Committee/Institutional Review Board. Relatedness to study vaccine was based on Investigator's discretion.
Time Frame: From Baseline (Day 0) up to 6 months after last vaccination (i.e., up to Month 7)
Population: Analysis was performed on the SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
Number analyzed (Participants) | 320 | 107 | 107 | 104
Participants
  SAE | 4 | 4 | 0 | 3
  SAE related to study vaccine | 0 | 2 | 0 | 0
  AESI | 0 | 0 | 0 | 0
  AESI related to study vaccine | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AE data were collected from Day 0 (post-vaccination 1) up to 28 days post any vaccination. SR data were collected within 7 days post any vaccination. SAE data were collected from Baseline (Day 0) up to 6 months after last vaccination (i.e., up to Month 7)
Description: Analysis was performed on SafAS. SR was an expected AR observed and reported under conditions (nature and onset) prelisted (i.e., solicited) in the protocol and CRB and considered as related to vaccination. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the CRB in terms of diagnosis and/or onset post-vaccination.
Arm/Group | Group 1 VRVg-2+HRIG | Group 2 Verorab+HRIG | Group 3 Imovax Rabies+HRIG | Group 4 VRVg-2
All-Cause Mortality (participants affected / at risk) | 0/320 | 0/107 | 0/107 | 0/104
Serious Adverse Events (participants affected / at risk) | 4/320 | 4/107 | 0/107 | 3/104
Other Adverse Events (participants affected / at risk) | 204/320 | 59/107 | 66/107 | 67/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 VRVg-2+HRIG (N=320) | Group 2 Verorab+HRIG (N=107) | Group 3 Imovax Rabies+HRIG (N=107) | Group 4 VRVg-2 (N=104)
General Physical Health Deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningioma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eating Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 VRVg-2+HRIG (N=320) | Group 2 Verorab+HRIG (N=107) | Group 3 Imovax Rabies+HRIG (N=107) | Group 4 VRVg-2 (N=104)
Fatigue (General disorders) | 3 (3) | 6 (6) | 1 (1) | 1 (1)
Injection Site Pain (General disorders) | 142 (337) | 37 (74) | 49 (118) | 44 (115)
Malaise (General disorders) | 34 (50) | 13 (15) | 14 (17) | 13 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 118 (221) | 37 (58) | 38 (71) | 34 (75) — Myalgia events that occurred after 7 days post-vaccination were considered as unsolicited AE.
Headache (Nervous system disorders) | 113 (173) | 35 (62) | 41 (59) | 40 (73) — Headache events that occurred after 7 days post-vaccination were considered as unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT03965962/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT03965962/SAP_001.pdf